CLINICAL TRIAL: NCT05296317
Title: Evaluation and Modeling of the Effect of G-CSF on the Evolution of Polynuclear Neutrophils During Dense Dose Epirubicin-Cyclophosphamide Regeneration
Acronym: EMEG-ECDD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-A01407-34
Record Dates: First submitted 2022-01-24; First posted 2022-03-25 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Localized Breast Cancer
Keywords: breast cancer; G-CSF; Epirubicin-cyclophosphamide dose-dense
MeSH Terms: conditions — Breast Neoplasms | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; Lenograstim; pegfilgrastim

STUDY DESIGN:
Intervention Model Description: Patients will be randomized :
  * Either to a peg-G-CSF arm (with administration of peg-G-CSF on D2)
  * Either to a G-CSF arm (with administration from D4 to D7 or D8). Blood samplig will be taken at D1, D4, D8 and D14 for each arm.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 : Dense dose epirubicin-cyclophosphamide chemotherapy with administration of G-CSF (Experimental): 2 cycles of chemotherapy with administration of G-CSF (filgrastim or lenograstim) on D2, D4 to D7 or D8..
  Realization of blood sampling at D1, D4, D8 and D14
  Interventions: Drug: Dense dose epirubicin-cyclophosphamide chemotherapy and G-CSF (filgrastim, lenograstim)
- Arm 2 : Dense dose epirubicin-cyclophosphamide chemotherapy with administration of peg-G-CSF (Experimental): 2 cycles of chemotherapy with administration of peg-G-CSF (pegfilgrastim) on D2.
  Realization of blood sampling at D1, D4, D8 and D14
  Interventions: Drug: Dense dose epirubicin-cyclophosphamide chemotherapy with administration of peg-G-CSF (pegfilgrastim)

INTERVENTIONS:
Drug: Dense dose epirubicin-cyclophosphamide chemotherapy and G-CSF (filgrastim, lenograstim) — - Arm 1: 2 cycles of chemotherapy with administration of G-CSF (filgrastim or lenograstim) on D2, D4 to D7 or D8..
  Realization of blood sampling at D1, D4, D8 and D14
  Arms: Arm 1 : Dense dose epirubicin-cyclophosphamide chemotherapy with administration of G-CSF
Drug: Dense dose epirubicin-cyclophosphamide chemotherapy with administration of peg-G-CSF (pegfilgrastim) — - Arm 2: 2 cycles of chemotherapy with administration of peg-G-CSF (pegfilgrastim) on D2.
  Realization of blood sampling at D1, D4, D8 and D14
  Arms: Arm 2 : Dense dose epirubicin-cyclophosphamide chemotherapy with administration of peg-G-CSF

SUMMARY:
Patients including of localized breast cancer will require chemotherapy treatment with epirubicin - cyclophosphamide (EC) followed by treatment with docetaxel or paclitaxel. In addition to this chemotherapy, the investigator will prescribe injections of granulocyte growth factors (G-CSF), to stimulate the growth of white blood cells. Patients will be randomized to either a peg-G-CSF arm or a G-CSF arm, prescribed at different times.

The aim is to determine whether one of the two treatment regimens best limits the risk of a decrease in white blood cells

DETAILED DESCRIPTION:
For this tudy : patients will be randomized to either :

* with administration of peg-G-CSF (administration on D2)
* with administration of G-CSF (administration on D4 to D7 or D8)

This study aims to model the effect of exogenous G-CSF for the evolution of polymorphonuclear neutrophils as a function of time and to explain the pharmacodynamic variability during the administration of chemotherapy such as EC-dense dose administered as an adjuvant or neo-adjuvant in patients treated for localized breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Patient over 18 years old
* Patient with histologically documented, non-metastatic breast cancer who must receive dense dose Epirubicin-Cyclophosphamide (EC) type treatment as part of neoadjuvant or adjuvant treatment
* Patient to receive granulocyte growth factors (G-CSF or peg-G-CSF) as a preventive measure from the first cycle
* Neutrophils > 1,500 /mm3; platelets > 100,000 /mm3
* Written informed consent, dated and signed
* For patients of childbearing age, effective means of contraception during treatment and up to 3 months after stopping treatment

Exclusion Criteria:

* Patient with a contraindication to treatment with anthracyclines
* Patient already undergoing treatment with EC dense dose
* Patient with a contraindication to treatment with G-CSF such as hypersensitivity to the active ingredient or to one of the excipients
* Pregnant or breastfeeding women
* Patient under guardianship or curatorship or subject to a protection regime for adults
* Patient not affiliated to a social security scheme (beneficiary or beneficiary)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — First inclusion criterion : Women
Enrollment: 100 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2025-09-02 (Estimated); Study Completion 2025-10-02 (Estimated)

PRIMARY OUTCOMES:
Variation of Neutrophils concentration in patient treated with G-CSF or peg-G-CSF | Day 4
  Variation of Neutrophils concentration will be assess by blood count formula performed during the 2 first cycle of Epirubicin-cyclophosphamide treatment.
Variation of Neutrophils concentration in patient treated with G-CSF or peg-G-CSF | Day 8
  Variation of Neutrophils concentration will be assess by blood count formula performed during the 2 first cycle of Epirubicin-cyclophosphamide treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Georges François Leclerc (CGFL), Dijon, Bourgogne-Franche-Comté, France